CLINICAL TRIAL: NCT02817815
Title: Atrial Fibrillation and Characterization of Blood Platelet
Acronym: FAPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure and non-replacement of the person in charge of the biological examinations specific to research carried out within the LIRYC IHU.
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2015/21
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation, blood platelet
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Active Comparator): Volunteers
  Interventions: Device: Electrocardiogram (ECG); Biological: Blood sampling from the cephalic vein
- Group 2 (Experimental): Paroxysmal AF patients in sinus rhythm the day of inclusion
  Interventions: Biological: Blood sampling from the femoral vein; Biological: First blood sampling from left atrium; Procedure: Atrial stimulation; Biological: Second blood sampling from left atrium
- Group 3 (Experimental): Paroxysmal AF patients in atrial fibrillation the day of inclusion
  Interventions: Biological: Blood sampling from the femoral vein; Biological: First blood sampling from left atrium
- Group 4 (Experimental): Persistent AF patients in sinus rhythm the day of inclusion
  Interventions: Biological: Blood sampling from the femoral vein; Biological: First blood sampling from left atrium; Procedure: Atrial stimulation; Biological: Second blood sampling from left atrium
- Group 5 (Experimental): Persistent AF patients in atrial fibrillation the day of inclusion
  Interventions: Biological: Blood sampling from the femoral vein; Biological: First blood sampling from left atrium

INTERVENTIONS:
Device: Electrocardiogram (ECG)
  Arms: Group 1
Biological: Blood sampling from the cephalic vein
  Arms: Group 1
Biological: Blood sampling from the femoral vein — Blood sampling will be done during radiofrequency ablation of AF procedure, after the introduction of catheter
  Arms: Group 2; Group 3; Group 4; Group 5
Biological: First blood sampling from left atrium — Blood sampling will be done during radiofrequency ablation of AF procedure, after transeptal punction
  Arms: Group 2; Group 3; Group 4; Group 5
Procedure: Atrial stimulation — Patients will receive atrial stimulation with the catheter positioned in the coronary sinus to induce AF
  Arms: Group 2; Group 4
Biological: Second blood sampling from left atrium — After 20min of continuous AF, a blood sampling from left atrium will be done
  Arms: Group 2; Group 4

SUMMARY:
Arterial thromboembolism constitutes a major risk of atrial fibrillation (AF) requiring antithrombotic therapy. Platelets and microparticles (MPs) are important for hemostasis and thrombosis, their role during AF is not well known. The principal objective of this study is to compare morphologic, functional and proteomics characteristics of blood platelet between AF patients and healthy volunteers.

DETAILED DESCRIPTION:
AF is associated with decreased quality of life and an increased risk of thromboembolic events. AF is the leading cause of embolic stroke. Identification of factors that may influence blood coagulability in these patients could better identify therapeutic targets to optimize anticoagulation. Platelets play a major role in the coagulation process, their study may provide valuable information. Moreover microparticles from platelet activation are known to have pathophysiological effects including effects on thrombosis and inhibition of fibrinolysis. It has also been shown that the microparticles have a role in endothelial dysfunction and generation of inflammatory condition which are associated with atrial fibrillation.

Investigators propose in this project, a comparative study between AF patients and healthy volunteers. Complete characterization of platelet (morphology, platelet function, platelet proteome) and microparticles levels will be perform. Different site blood sampling (systemic or cardiac) will be done in patients during their ablation procedure. Patients will be followed during their hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: valid for all groups

  * Age superior or equal to 18 years old, both genders.
  * Patient affiliated or recipient of a social welfare regimen.
  * Patient's write agreement for study participation after reading information note
* Inclusion Criteria: specific for groups

Group 1:

* Volunteers without heart disease.
* Volunteers who never had AF and not in AF the day of inclusion. Group 2
* Patient suffering of paroxysmal atrial fibrillation since at least 6 month and addressed for primo ablation of atrial fibrillation.
* Patient in sinus rhythm the day of inclusion. Group 3
* Patient suffering of paroxysmal atrial fibrillation since at least 6 month and addressed for primo ablation of atrial fibrillation.
* Patient in atrial fibrillation the day of inclusion Group 4
* Patient suffering of persistent atrial fibrillation since at least 6 month and addressed for primo ablation of atrial fibrillation.
* Patient in sinus rhythm the day of inclusion. Group 5
* Patient suffering of persistent atrial fibrillation since at least 6 month and addressed for primo ablation of atrial fibrillation.
* Patient in atrial fibrillation the day of inclusion

Exclusion Criteria:

* Age <18 years.
* Active smoker (> 10 cigarettes/days)
* Pregnant woman or breastfeeding women or not receiving effective contraception.
* Volunteer participating in another interventional study requiring taking drug.
* Volunteer having taken antinflammatory, platelet anti-aggregant or calcium-channel blocker drugs within 8 days prior to inclusion
* Valvular heart diseases.
* Chronic inflammatory diseases.
* Cardiovascular event or stroke within 3 month prior to inclusion
* Uncontrolled hypertension
* Chronic hepatic or renal diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Measure of maximal aggregation level (expressed in aggregation percentage) after ex vivo stimulation by Adenosine Di-Phosphate (ADP), arachidonic acid, ristocetin, collagen and Thrombin Receptor Activating Peptide (TRAP-6mers) | Day 1
  Aggregation percentage is measured by the method of light transmission aggregometry
Measure of maximal disaggregation level (expressed in disaggregation percentage) | Day 1
  Disaggregation percentage is measured by the method of light transmission aggregometry
Measure of platelet volume mean | Day 1
Assessment of the Platelet morphology (shape change) | Day 1
Assessment of the modification of the membrane receptor expression modification | Day 1
Identification of platelet proteins differentially expressed between groups | Day 1

SECONDARY OUTCOMES:
Measure of Tissue Factor (TF) dependent microparticles level | Day 1
Measure of fibrinolytic microparticles level | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Electrophysiologie et de stimulation cardiaque / LIRYC - Hôpital Cardiologique du Haut Lévêque, Pessac, France